CLINICAL TRIAL: NCT00544102
Title: Insulin Resistance and Atherosclerosis in a Sample of Women With Systemic Lupus Erythematosus
Brief Title: Insulin Resistance and Atherosclerosis in Women With Lupus
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080008; 08-AR-0008
Record Dates: First submitted 2007-10-14; First posted 2007-10-16 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2017-09-07

CONDITIONS: Systemic Lupus Erythematosus; Insulin Resistance; Atherosclerosis
Keywords: Insulin Resistance; Systemic Lupus Erythematosus; Atherosclerosis; Lupus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Insulin Resistance; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
This study will test the effects of insulin resistance on atherosclerosis (hardening of the arteries) in women who have systemic lupus erythematosus, more commonly known as lupus. Women with lupus have a higher chance of developing atherosclerosis than the general population, and as a result are more susceptible to heart attack and stroke. Insulin resistance is a particular risk factor for atherosclerosis, and recent small studies have shown that insulin resistance is more common in lupus patients than in those without lupus. The study will consist of a series of tests designed to assess whether there is an association between insulin resistance and atherosclerosis in women with lupus. This research may lead to further studies on possible treatments to reduce the risk of heart disease in lupus patients.

Volunteers must be women between 30 and 55 years of age who were diagnosed with lupus within five or more years prior to the study. Volunteers who have kidney failure, diabetes, or existing atherosclerosis will be excluded from the study, as will volunteers who have had pulse steroid therapy within four weeks of the testing or who have been pregnant within one year of the testing.

Participants will undergo the following procedures on an outpatient basis:

* Blood and urine tests for research purposes.
* Electrocardiogram (EKG) to test the general health of the heart.
* Oral glucose tolerance test to measure blood glucose and insulin levels. This test is commonly used to diagnose diabetes and pre-diabetic insulin resistance.
* Cardiac multidetector computed tomography (MDCT) to determine the amount of calcium present in coronary arteries. This test is used to diagnose atherosclerosis.
* Carotid artery ultrasound to show the speed of blood flow through the carotid arteries. This test will show abnormalities and/or blockages in the carotid arteries.
* Abdominal ultrasound to determine if the participant has hepatic steatosis ( fatty liver ), which is often found in individuals with insulin resistance and diabetes.
* Carotid artery magnetic resonance imaging/angiogram (MRI/MRA) to measure the thickness of blood vessels. This test is used to diagnose atherosclerosis.
* Abdominal MRI to estimate abdominal fat.

Volunteers may be asked to participate in an MRI/MRA study to evaluate the arteries of the heart. This test is optional and not required by the insulin resistance/atherosclerosis study. The entire series of procedures will require one to three visits to complete.

DETAILED DESCRIPTION:
Women with lupus have a five- to ten-fold increased risk of coronary heart disease compared to the general population. Several decades ago, when women with lupus died shortly after developing the disease, their deaths were attributed to previously undiagnosed and untreated active lupus. But when they died years after their diagnosis of lupus, their deaths were attributed to complications of atherosclerosis (hardening of the arteries). Similar to lupus, atherosclerosis is considered an inflammatory disease. Inflammation plays a major role in atherosclerosis, which results when fatty deposits, cholesterol and other materials accumulate in the blood vessels.

The combination of atherosclerosis and lupus greatly increases the risk of cardiovascular disease among women. Research has identified many factors that contribute to the risk of atherosclerosis in people with lupus. These include high blood pressure and abnormal cholesterol levels, chronic inflammation, antibodies that attack proteins that regulate the blood vessels, and some medications used to treat lupus.

In the general population, diabetes is an important risk factor for atherosclerosis. A silent condition called insulin resistance can lead to diabetes and has been associated with atherosclerosis in populations that do not have lupus. Recent studies have shown people with lupus are more likely to have insulin resistance than those without the disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Women 30-55 years of age.
* Must give written informed consent prior to entry in the protocol.
* Must fulfill at least 4 of the classification criteria for SLE as defined by the American College of Rheumatology.
* Diagnosis of SLE made 5 or more years prior to study participation.

EXCLUSION CRITERIA:

* Pregnancy within one year of study participation. Women of childbearing potential are required to have a negative pregnancy test at screening.
* Previous diagnosis of Type 1 or 2 diabetes mellitus.
* History of cerebrovascular accident (CVA: presence of irreversible or partially reversible motor and/or sensory deficits of sudden or recent onset on the basis of vascular occlusion or insufficiency, complete, incomplete or in evolution, persisting greater than 24 hours or lasting less than 24 hours with an anatomic correlate).
* Previous diagnosis of peripheral vascular disease (PVD: presence of arterial claudication [pain in the muscles of the upper or lower extremities, induced by exercise and relieved by rest, with absent pulses and/or confirmed by Doppler flow studies and/or angiography] lasting greater than 6 months and/or evidence of gangrene or significant tissue (digit or limb) loss not attributable to Raynaud s phenomenon).
* Therapy with pulse methylprednisolone or pulse prednisone within 4 weeks of study participation.
* Initiation or change in dosage of antilipemic agents within the preceding six weeks.
* Any active viral or bacterial infection
* Significant concurrent medical condition that, in the opinion of the Principal Investigator, could affect the patient s ability to tolerate or complete the study.
* Clinical coronary artery disease (CAD) defined as: history of MI and/or definite or classic angina (substernal chest discomfort provoked by exertion or emotion and relieved by rest or nitroglycerine), and/or conclusive evidence of MI on ECG
* Renal failure defined as hemodialysis-dependant, or calculated GFR less than or equal to 30 mL/minute (calculated by the MDRD 4 variable formula).

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-10-11; Study Completion 2017-09-07

PRIMARY OUTCOMES:
Correlation of insulin resistance with coronary atherosclerosis

SECONDARY OUTCOMES:
Prevalance of insulin resistance and impaired glucose tolerance in SLE prevalence of atherosclerosis via coronary artery measurements, correlation of insulin resistance and potential bio-markers SHBG and retinal binding protein

CONTACTS AND LOCATIONS:
Overall Officials: Sarfaraz A Hasni, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Manzi S, Meilahn EN, Rairie JE, Conte CG, Medsger TA Jr, Jansen-McWilliams L, D'Agostino RB, Kuller LH. Age-specific incidence rates of myocardial infarction and angina in women with systemic lupus erythematosus: comparison with the Framingham Study. Am J Epidemiol. 1997 Mar 1;145(5):408-15. doi: 10.1093/oxfordjournals.aje.a009122. PMID 9048514
- [Background] Doria A, Shoenfeld Y, Wu R, Gambari PF, Puato M, Ghirardello A, Gilburd B, Corbanese S, Patnaik M, Zampieri S, Peter JB, Favaretto E, Iaccarino L, Sherer Y, Todesco S, Pauletto P. Risk factors for subclinical atherosclerosis in a prospective cohort of patients with systemic lupus erythematosus. Ann Rheum Dis. 2003 Nov;62(11):1071-7. doi: 10.1136/ard.62.11.1071. PMID 14583570
- [Background] Bruce IN, Burns RJ, Gladman DD, Urowitz MB. Single photon emission computed tomography dual isotope myocardial perfusion imaging in women with systemic lupus erythematosus. I. Prevalence and distribution of abnormalities. J Rheumatol. 2000 Oct;27(10):2372-7. PMID 11036832